CLINICAL TRIAL: NCT01858389
Title: Phase 2 Open Label Trial Of Oral Intermittent Dacomitinib In Patients With Advanced Nsclc
Brief Title: A Study Of Dacomitinib (PF-00299804) In Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A7471047
Record Dates: First submitted 2013-05-06; First posted 2013-05-21 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; T790M mutation. dacomitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Patients with NSCLC whose tumor has a documented T790M mutation in exon 20 of the Epidermal Growth Factor Receptor.
  Interventions: Drug: Dacomitinib
- Cohort B (Experimental): Patients with NSCLC. No requirement of a specific molecular signature, but excluding known T790M mutations.
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Dacomitinib 45 mg every 12 hours Days 1-4 of the first week, and then 60 mg every 12 hours Days 1-4 of each 2-week cycle thereafter. The dose of dacomitinib for patients in Cohort A may be further escalated in increments of 15 mg.
  Arms: Cohort A
Drug: Dacomitinib — Dacomitinib 45 mg every 12 hours Days 1-4 of the first week, and then 60 mg every 12 hours Days 1-4 of each 2-week cycle thereafter.
  Arms: Cohort B

SUMMARY:
This is a Phase 2 study of oral dacomitinib given every 12 hours over days 1-4 of each two-week cycle to patients with Non-small cell lung cancer. The study includes two groups of patients, those whose tumor has a documented T790M mutation, and those without this mutation. All patients will receive repeated cycles of dacomitinib until disease progression, occurrence of unacceptable toxicity, or other withdrawal criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of histologically confirmed, advanced NSCLC (stage IIIB/IV).
* Evidence of T790M mutation to enroll in Cohort A.
* Evidence of measurable disease by radiographic technique.
* Adequate organ function.

Exclusion Criteria:

* Patients with T790M mutation who stopped any prior EGFR-directed therapy without evidence of disease progression.
* Symptomatic brain metastases.
* Uncontrolled or significant cardiovascular disease.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (12):
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Georgetown University Hospital-Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Georgetown University Medical Center Department of Pharmacy, Research, Washington D.C., District of Columbia
  - Memorial Sloan-Kettering Cancer Center-Rockefeller Outpatient Pavilion, New York, New York
  - Investigational Drug Service, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center-Simmons Cancer Center Pharmacy, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Southwestern University Hospital - William P. Clements, Jr., Dallas, Texas
  - UT Southwestern University Hospital - Zale Lipshy, Dallas, Texas
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Tan W, Giri N, Quinn S, Wilner K, Parivar K. Evaluation of the potential effect of dacomitinib, an EGFR tyrosine kinase inhibitor, on ECG parameters in patients with advanced non-small cell lung cancer. Invest New Drugs. 2020 Jun;38(3):874-884. doi: 10.1007/s10637-019-00887-0. Epub 2019 Dec 19. PMID 31858327
- [Derived] Yu HA, Ahn MJ, Cho BC, Gerber DE, Natale RB, Socinski MA, Giri N, Quinn S, Sbar E, Zhang H, Giaccone G. Phase 2 study of intermittent pulse dacomitinib in patients with advanced non-small cell lung cancers. Lung Cancer. 2017 Oct;112:195-199. doi: 10.1016/j.lungcan.2017.08.017. Epub 2017 Aug 23. PMID 29191595
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471047&StudyName=A%20Study%20Of%20Dacomitinib%20%28PF-00299804%29%20In%20Patients%20With%20Advanced%20Non-Small%20Cell%20Lung%20Cancer%20%0A

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 41 participants enrolled in the study, 38 (16 with T790M mutation and 22 without T790M mutation) received study drug. Three of the enrolled participants without known T790M mutation did not receive treatment.
Groups:
- Dacomitinib, 45/60 mg, With T790M Mutation: Participants with documented T790M mutation in exon 20 of epidermal growth factor receptor received dacomitinib, 45 mg, every 12 hours for 6 doses over Days 1-4 of a 1-week lead-in cycle. Following the lead-in cycle, all participants received dacomitinib, 60 mg, every 12 hours for 6 doses over Days 1-4 of each subsequent 2-week cycle. Dose could be escalated beyond 60 mg after consultation with and approval of the sponsor.
- Dacomitinib, 45/60 mg, Without T790M Mutation: Participants with no known T790M mutation received dacomitinib, 45 mg, every 12 hours for 6 doses over Days 1-4 of a 1-week lead-in cycle. Following the lead-in cycle, all participants received dacomitinib, 60 mg, every 12 hours for 6 doses over Days 1-4 of each subsequent 2-week cycle.
Period: Overall Study
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation | Dacomitinib, 45/60 mg, Without T790M Mutation
Started | 16 (Enrolled) | 25 (Enrolled)
Received Treatment | 16 | 22
Completed | 0 | 0
Not Completed | 16 | 25
Not completed — Death | 1 | 3
Not completed — Study terminated by sponsor | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive disease | 10 | 11
Not completed — Other | 2 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Did not receive treatment | 0 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation | Dacomitinib, 45/60 mg, Without T790M Mutation | Total
Number analyzed (Participants) | 16 | 22 | 38
Age, Customized [Number; unit: Participants]
  Younger than 18 years | 0 | 0 | 0
  Between 18 and 44 years | 2 | 0 | 2
  Between 45 and 64 years | 9 | 13 | 22
  65 years and older | 5 | 9 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 4 | 10 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 6 | 9 | 15
  Black or African American | 2 | 2 | 4
  Asian | 7 | 10 | 17
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) in Participants With T790M Mutation
Description: BOR was best response from start of treatment until disease progression, according to the RECIST,v1.1. CR=disappearance of all preexisting lesions except nodal disease, with all nodal lesions decreased to normal size (short axis <10 mm) and no appearance of new unequivocal malignant lesions. PR= ≥30% decrease from baseline of sum of diameters of all target lesions with no unequivocal progression of preexisting non-target lesions or appearance of new lesions. CR and PR were confirmed on a follow-up imaging assessment ≥4 weeks after the initial response documentation. Progression= ≥20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions or appearance of any new unequivocal malignant lesions. Stable disease=not qualify for CR, PR or progression. BOR was analyzed only for participants with T790M mutation according to the primary study objective.
Time Frame: From baseline until disease progression, up to 61 weeks.
Population: All enrolled participants with T790M mutation
Measure: Number; unit: Participants
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation
Number analyzed (Participants) | 16
Participants
  Complete response (CR) | 0
  Partial response (PR) | 1
  Stable disease/no response | 7
  Objective progression | 6
  Indeterminate | 2

2. Secondary Outcome: Disease Control Rate (DCR) for Participants With T790M Mutation
Description: DCR was calculated as the percentage of participants with an objective response (CR or PR) or stable disease, based on the RECIST, v1.1, relative to the total number of participants enrolled in the cohort. If baseline tumor assessment was inadequate for a participant, and the participant could not be assessed for RECIST responses and had no objective status of stable disease documented at least 6 weeks after the start date and before the progression, the participant was only counted in the denominator. CR=disappearance of all preexisting lesions except nodal disease, with all nodal lesions decreased to normal size (short axis <10 mm) and no appearance of new unequivocal malignant lesions. PR= ≥30% decrease from baseline of sum of diameters of all target lesions with no unequivocal progression of preexisting non-target lesions or appearance of new lesions. DCR was analyzed only for participants with T790M mutation according to the study objective.
Time Frame: From baseline to baseline to disease progression, up to 61 weeks.
Population: All enrolled participants with T790M mutation
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation
Number analyzed (Participants) | 16
Percentage of participants | 50 [24.7 to 75.3]

3. Secondary Outcome: Duration of Response in Participants With T790M Mutation
Description: Duration of response was defined as the time from first documentation of response (CR or PR, whichever occurred first) to the date of disease progression or to death due to any cause, whichever occurred first. CR and PR were defined using RECIST, v1.1. CR=disappearance of all preexisting lesions except nodal disease, with all nodal lesions decreased to normal size (short axis <10 mm) and no appearance of new unequivocal malignant lesions. PR= ≥30% decrease from baseline of sum of diameters of all target lesions with no unequivocal progression of preexisting non-target lesions or appearance of new lesions. CR and PR were confirmed on a follow-up imaging assessment ≥4 weeks after the initial response documentation. DR was only calculated and summarized for the subgroup of participants with an objective tumor response in the cohort of participants with T790M mutation.
Time Frame: From baseline to date of disease progression or death, up to 61 weeks.
Population: All enrolled participants with T790M mutation status who had an objective tumor response (complete or partial response)
Measure: Number; unit: Months
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation
Number analyzed (Participants) | 1
Months | 2.83

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the date of first dosing of dacomitinib to the date of disease progression by RECIST v1.1, per the investigators' assessment, or death due to any cause, whichever occurred first. Objective progression= ≥20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions or appearance of any new unequivocal malignant lesions.
Time Frame: From baseline to disease progression or death, up to 61 weeks.
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation | Dacomitinib, 45/60 mg, Without T790M Mutation
Number analyzed (Participants) | 16 | 25
Months | 2.3 [1.4 to 4.4] | 1.6 [1.0 to 3.3]

5. Secondary Outcome: Progression-free Survival at 4 Months
Description: Progression-free survival at 4 months was defined as the percentage of participants who were alive without disease progression at 4 months relative to all participants enrolled. Disease progression was defined by RECIST v1.1. Objective progression= ≥20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions or appearance of any new unequivocal malignant lesions.
Time Frame: Month 4
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation | Dacomitinib, 45/60 mg, Without T790M Mutation
Number analyzed (Participants) | 16 | 25
Percentage of participants | 37.5 [15.4 to 59.8] | 25.3 [8.6 to 46.2]

6. Primary Outcome: Objective Response Rate (ORR) in Participants With T790M Mutation
Description: ORR was calculated as the percentage of participants with a confirmed CR or PR relative to the total number of participants enrolled. Response Evaluation Criteria in Solid Tumors (RECIST), version (v) 1.1 were used to define CR and PR. CR=disappearance of all preexisting lesions except nodal disease, with all nodal lesions decreased to normal size (short axis <10 mm) and no appearance of new unequivocal malignant lesions. PR= ≥30% decrease from baseline of sum of diameters of all target lesions with no unequivocal progression of preexisting non-target lesions or appearance of new lesions. CR and PR were confirmed on a follow-up imaging assessment ≥4 weeks after the initial response documentation. ORR was analyzed only for participants with T790M mutation according to the primary study objective.
Time Frame: From baseline to disease progression, up to 61 weeks.
Population: All enrolled participants with T90M mutation
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation
Number analyzed (Participants) | 16
Percentage of participants | 6.3 [0.2 to 30.2]

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Dacomitinib and PF-05199265
Description: Cmax was observed directly from data. Whole blood for pharmacokinetic analysis was collected immediately after completion of electrocardiograms, blood pressure, and pulse rate.
Time Frame: Pre-dose (hour 0), 2, 4, 6, 8, and 10 hours post-dose on Day 4, Cycle 0.
Population: All participants who received at least 1 dose of study drug and who had at least 1 measured plasma concentration of dacomitinib or its major circulating metabolite PF 05199265.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dacomitinib, 45 mg: Participants received a 1-week lead-in cycle of dacomitinib, 45 mg, every 12 hours for 6 doses on Days 1-4.
Arm/Group | Dacomitinib, 45 mg
Number analyzed (Participants) | 37
ng/mL
  Dacomitnib | 96.76 (37.510)
  PF-05199265 (Dacomitnib metabolite) | 8.45 (12.648)

8. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Dacomitinib and PF-05199265
Description: Tmax was observed directly from data as time of first occurrence. Whole blood for pharmacokinetic analysis was collected immediately after completion of electrocardiograms, blood pressure, and pulse rate.
Time Frame: Pre-dose (hour 0), 2, 4, 6, 8, and 10 hours post-dose on Day 4, Cycle 0.
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Dacomitinib, 45 mg
Number analyzed (Participants) | 37
Hours
  Dacomitinib | 6.07 [1.3 to 10.9]
  PF-05199265 | 5.58 [0.0 to 11.0]

9. Secondary Outcome: Changes From Time-matched Baseline in Adjusted Fridericia Corrected QT Interval (QTcF) on Echocardiogram (ECG)
Description: ECGs recorded on Day 1 of Cycle 0 were used as baseline. For the ECGs assessments, the following directions were followed by the ECG central laboratory: Blinding of ECG readers to treatment, time, and day identifiers. Review of ECGs from a particular participant was performed by a single reader. Prespecification of the lead for internal measurements. Baseline and on-treatment ECG assessments were based on the same lead.
Time Frame: From Baseline to Cycle 0, Day 4
Population: All participants who received all scheduled doses of dacomitinib and had all ECGs performed on Days 1-4 of Cycle 0 (n=number evaluable)
Measure: Mean (90% Confidence Interval); unit: msecs
Groups:
- Dacomitinib, 45/60 mg: Participants received a 1-week lead-in cycle of dacomitinib, 45 mg, every 12 hours for 6 doses on Days 1-4. Following the lead-in cycle, all participants received intermittent dacomitinib, 60 mg, administered every 12 hours for 6 doses at the beginning of each 2-week cycle.
Arm/Group | Dacomitinib, 45/60 mg
Number analyzed (Participants) | 32
msecs
  QTcF Interval Cycle 0, Day 4: Hour 0 | 1.7 [-2.33 to 5.64]
  QTcF Interval Cycle 0, Day 4: Hour 2 | 4.4 [1.85 to 6.97]
  QTcF Interval Cycle 0, Day 4: Hour 4 | 0.4 [-3.89 to 4.64]
  QTcF Interval Cycle 0, Day 4: Hour 6 (n=31) | -0.4 [-3.98 to 3.14]
  QTcF Interval Cycle 0, Day 4: Hour 8 (n=31) | 0.1 [-2.43 to 2.63]
  QTcF Interval Cycle 0, Day 4: Hour 10 (n=31) | 0.5 [-2.58 to 3.68]

ADVERSE EVENTS:
Arm/Group | Dacomitinib, 45/60 mg, With T790M Mutation | Dacomitinib, 45/60 mg, Without T790M Mutation
Serious Adverse Events (participants affected / at risk) | 7/16 | 8/22
Other Adverse Events (participants affected / at risk) | 16/16 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib, 45/60 mg, With T790M Mutation (N=16) | Dacomitinib, 45/60 mg, Without T790M Mutation (N=22)
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib, 45/60 mg, With T790M Mutation (N=16) | Dacomitinib, 45/60 mg, Without T790M Mutation (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 1
Eye irritation (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 14 | 16
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 9
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 2 | 3
Chest pain (General disorders) | 1 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 7
Gait disturbance (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 2
Local swelling (General disorders) | 1 | 0
Mass (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 3
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0
Xerosis (General disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Carbuncle (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Ear infection fungal (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 4 | 7
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase decreased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0
Human chorionic gonadotropin increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 7
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 8 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.